CLINICAL TRIAL: NCT05442606
Title: Effect of Adding Physiotherapy Program to the Conservative Medical Therapy on Quality of Life and Pain Threshold in Chronic Rhinosinusitis Patients: A Prospective Randomized Controlled Trial
Brief Title: Physiotherapy Protocol in Treating Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Jouf University (Other)
Responsible Party: Principal Investigator, Khaled Z. Fouda, Associate Professor of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-13-S-071(071)
Record Dates: First submitted 2022-06-26; First posted 2022-07-05 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Rhinosinusitis
Keywords: Rhinosinusitis; ultrasound therapy; quality of life; pain threshold; manual therapy
MeSH Terms: conditions — Rhinosinusitis | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative medical therapy (No Intervention): Patients in this group received only medication prescribed by an Ear, Nose and Throat specialist.
- Medication and Physiotherapy program (Experimental): Patients in this group received medication prescribed by an Ear, Nose and Throat specialist, in addition to integrated Physiotherapy program
  Interventions: Other: Ultrasound Therapy; Other: Manual Drainage Techniques; Other: Self Sinus Massage Technique

INTERVENTIONS:
Other: Ultrasound Therapy — Using an Enraf Nonius Sonoplus 490 from the Netherlands, the patients were asked to lie supine while the therapist stood at the level of the patient's head. The patients received pulsed (duty cycle 50%) US therapy with intensities of 1 and 0.5 W/cm2 for maxillary and frontal sinus, respectively, and a collimating beam frequency of 1MHz. To deliver US to the treatment area, a small probe US applicator (0.8 cm2) with an effective radiating area (ERA) of 0.6 cm2 and a beam non-uniformity ratio (BNR) of 6:1 was used. The skin around the cheeks was used for the maxillary sinus and the forehead for the frontal sinus. Between the applicator and the skin, ultrasound transmission gel was employed, and a full contact technique in slow circular motion was used for 5 minutes over the maxillary sinuses and 4 minutes over the frontal sinuses on each pair of sinuses
  Arms: Medication and Physiotherapy program
Other: Manual Drainage Techniques — Manual Drainage Techniques for the frontal and maxillary sinuses
  Arms: Medication and Physiotherapy program
Other: Self Sinus Massage Technique — Patients will also encouraged to self-massage their frontal and maxillary sinuses while resting supine
  Arms: Medication and Physiotherapy program

SUMMARY:
This study aims to investigate the effect of adding of integrated physiotherapy program to the conservative medical therapy on quality of life and pressure pain threshold (PPT) in chronic rhinosinusitis patients. Patients in this study will be randomly assigned into 2 groups. Group A (control group) will receive conservative medical treatment only which prescribed by Ear, Nose and Throat (ENT) specialist, while group B (experimental group) will receive the conservative medical treatment prescribed by ENT specialist in addition to physiotherapy program. Quality of Life (QoL) will be evaluated by Rhinosinusitis Disability Index (RSDI) and PPT will be evaluated by digital algometer at the baseline and immediately after the end of tenth session of treatment for both groups.

DETAILED DESCRIPTION:
Sixty-eight patients will be recruited for this study from Al-Qurayyat General Hospital in Al-Jouf Region, Saudi Arabia, with the following inclusion criteria: patients of both sexes, aged from 30 to 50 years, diagnosed by ENT specialist, with chronic rhinosinusitis with a history of 3 months or longer. The patients will be allocated into two equal groups at random (n = 34). Group A (control group) will receive medication only which prescribed by ENT specialist. Group B (experimental group) will receive prescribed medication by ENT specialist in addition to physiotherapy program which consists of: Ultrasound Therapy: The patients will receive pulsed (duty cycle 50%) US therapy with an intensity of 1 and 0.5 W/cm2 for maxillary and frontal sinus, respectively, with a frequency of 1MHz collimating beam. The small probe US applicator (0.8 cm2) with effective radiating area (ERA) equal 0.6 cm2 and beam non-uniformity ratio (BNR) equal 6:1 will be used to deliver US to the treatment area. The area of US application will be the skin over the cheeks for maxillary sinus and forehead for the frontal sinus. Ultrasound transmission gel will be used between the applicator and the skin, full contact technique in slow circular motion will be used for the duration of 5 minutes over the maxillary sinuses and 4 minutes over the frontal sinuses on each pair of sinuses. Manual Drainage Techniques: for the frontal and maxillary sinuses. Self Massaging Technique: The patients will also advised to perform self-massaging for the frontal and maxillary sinuses from the supine lying position. A demonstration session will be used to provide patients in the experimental group with a full description of the manual therapy procedure before the beginning of the study. The physiotherapy program will be applied 3 times a week (day after day) for 12 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Aged from 30 to 50 years
* Cynically diagnosed by Ear, Nose, and Throat (ENT) specialist, with chronic rhinosinusitis with a history of more than 3 months, confirmed by clinical diagnostic criteria (more than or equal to two major symptoms or one major symptom (nasal obstruction, facial pain/pressure, postnasal drip and hyposmia) and two minor symptoms (headache, halitosis, fatigue, dental pain and ear pain) and also verified by Computed Tomography (CT) scan results .

Exclusion criteria:

* Having any tumors or cysts (as confirmed by CT scan)
* Nasal polyps
* Facial skin lesions or diseases or allergies of the face
* Pregnancy
* Metal implants in the face region
* Previous nasal surgical procedures
* Impaired thermal sensation (such as uncontrolled diabetes mellitus)
* Cognitive level impairment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Rhinosinusitis Disability Index (RSDI) | From baseline to 4 weeks after treatment (immediately after the completion of session 12)
  Arabic version of Rhinosinusitis Disability Index will be used to assess the change in quality of life

SECONDARY OUTCOMES:
Pressure pain threshold | From baseline to 4 weeks after treatment (immediately after the completion of session 12)
  Wagner FPX25 digital algometer will be used to assess the change in pressure pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Fouda, PhD, Principal Investigator — Associate Professor of Physical Therapy
Locations (1):
- Al Qurayyat General Hospital, Qurayyat, Jouf Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared including a summary of the results after the study completion date.
Supporting Information: Study Protocol
Time Frame: The dead time for IPD will be 30 June.2025
Access Criteria: will be uploaded on the official site of CTR
URL: https://www.e-arm.org/journal/view.php?doi=10.5535/arm.23058

REFERENCES:
- See also: Free Full Paper — https://www.e-arm.org/journal/view.php?doi=10.5535/arm.23058
- Available data/document: Full Paper — https://www.e-arm.org/journal/view.php?doi=10.5535/arm.23058